CLINICAL TRIAL: NCT06731101
Title: The Efficacy of Stellate Ganglion Block Versus Combined Oral Anticholinergic and Antidepressant Drugs on Treatment of Palmar Hyperhidrosis; A Randomized Comparative Study
Brief Title: Stellate Ganglion Block Versus Oral Medication in Treatment of Palmar Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Taha mohamed agmy, Atef Mohamed Mahmoud, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D401
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Palmar Hyperhidrosis
Keywords: Stellate ganglion block
MeSH Terms: interventions — Bupivacaine; Lidocaine; chlordiazepoxide, clidinium drug combination; Anti-Anxiety Agents

STUDY DESIGN:
Intervention Model Description: Compare two groups of Palmar hyperhidrosis one with injection Local anesthetic at stellate ganglion, the other will take oral medication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate ganglion block (Active Comparator): bupivacaine+ lidocaine + dexamethasone injection into stellate ganglion
  Interventions: Drug: Bupivacaine + Lidocaine +dexamethasone
- Drugs (Active Comparator): librax + tryptizole
  Interventions: Drug: Tryptizole + Librax

INTERVENTIONS:
Drug: Bupivacaine + Lidocaine +dexamethasone — Sonar guided block of Stellate Ganglion By Bupivacaine + Lidocaine
  Other Names: xylocaine or bupivacine; lidocaine or marcaine
  Arms: Stellate ganglion block
Drug: Tryptizole + Librax — Tryptizole + Librax
  Other Names: Anxiolytics
  Arms: Drugs

SUMMARY:
The aim of the study is to compare between ganglion block versus combined oral anticholinergic and antidepressant drugs on treatment of palmar hyperhidrosis

DETAILED DESCRIPTION:
Palmar hyperhidrosis is a medical condition characterized by excessive sweating specifically from the palms of the hands. This condition can significantly impact an individual's quality of life, leading to social embarrassment, anxiety, and difficulties in daily activities. It is classified as a type of primary hyperhidrosis, which means it occurs without an identifiable underlying medical cause (Solish et al., 2022).

The prevalence of palmar hyperhidrosis is estimated to affect about 1% to 3% of the population. Symptoms typically begin in childhood or adolescence, often becoming more pronounced during periods of hormonal changes such as puberty. The condition may run in families, suggesting a genetic predisposition (Wadhawa et al., 2019).

The underlying mechanism involves hyperactivity of the sympathetic nervous system, particularly affecting the eccrine sweat glands located in the palms (Kisielnicka et al., 2022).

Unlike normal sweating, which primarily serves thermoregulation (cooling the body), palmar hyperhidrosis is triggered by emotional stimuli such as stress or anxiety rather than heat. This inappropriate activation leads to excessive sweating that can occur even at rest (Schote et al., 2022).

Diagnosis is primarily clinical and based on patient history and visible signs of excessive sweating. Patients often report episodes that are bilateral and symmetrical, with cold and wet palms that may appear pale or blushed. The diagnosis does not typically require extensive testing unless secondary causes are suspected (Henning et al., 2021).

Treatment for palmar hyperhidrosis can be challenging due to varying degrees of severity and individual responses to therapies (Chudry, 2022).

Common treatment options include topical treatments as aluminum chloride hexahydrate which is considered one of the most effective topical treatments for palmar hyperhidrosis. It works by blocking sweat pores and reducing gland activity. Application involves using a concentrated solution on dry skin at night until symptoms improve, followed by maintenance therapy (Rahim et al., 2022).

Another option of treatment is iontophoresis; this technique uses electrical currents to temporarily block sweat gland function. It requires multiple sessions but can be effective for many patients (Nastase et al., 2024).

Botulinum toxin type A can be injected into affected areas to inhibit neurotransmitter release responsible for activating sweat glands. While effective, this treatment requires repeated injections every few months due to its temporary effects (Martina et al., 2021).

Anticholinergic drugs have been used but are often limited by side effects such as dry mouth and constipation at effective dosages (Wong et al., 2022).

The stellate ganglion block (SGB) is a nonsurgical treatment option for managing hyperhidrosis, particularly in cases where other treatments have failed. The stellate ganglion is a collection of nerves located in the neck that plays a crucial role in regulating sweat gland activity. By blocking these nerves, it is possible to reduce sweating in the affected areas (Deng et al., 2023).

The SGB works by injecting local anesthetics into the stellate ganglion, which interrupts the sympathetic nerve signals responsible for activating sweat glands. This procedure can be performed using ultrasound guidance to ensure accurate placement of the needle. The typical approach involves administering an anesthetic such as lidocaine or bupivacaine directly into the ganglion (Feigin et al., 2023).

Regarding surgical options; surgical sympathectomy is considered a last resort for severe cases where other treatments have failed. This procedure involves cutting nerves that trigger sweating but carries risks such as compensatory sweating in other body areas (Kuijpers et al., 2022).

Finally, palmar hyperhidrosis is a common yet often underreported condition that can severely affect individuals' lives due to its social implications and discomfort associated with excessive sweating. Treatment options vary widely in effectiveness and side effects, necessitating a tailored approach based on individual needs (Trettin et al., 2022).

ELIGIBILITY:
Inclusion criteria: -

1. Age from 20 to 45 years.
2. Both genders.
3. Exhibiting primary palmar hyperhidrosis. Exclusion criteria: -

1. An inability of patient to cooperate. 2. Known allergies to anticholinergic or antidepressant drugs.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Secretions | 3 months
  i.e. presence/absence of hyperhidrosis

SECONDARY OUTCOMES:
Compensatory hyperhidrosis | 1 ]week
  Increase secretions in other side

CONTACTS AND LOCATIONS:
Overall Officials: Atef M Khalil, professor, Principal Investigator — Fayoum University
Locations (1):
- Taha mohamed agmy, Al Fayyum, Egypt